CLINICAL TRIAL: NCT05477199
Title: Cognitive Behavioral Principles-based Treatment Program for Patients With Post COVID-19 Syndrome
Brief Title: Physiotherapy in Post COVID-19 Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DF0098UG
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2022-07

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral principles-based treatment program group (Experimental)
  Interventions: Other: Cognitive behavioral principles-based treatment program
- Control group (Active Comparator)
  Interventions: Other: Control intervention

INTERVENTIONS:
Other: Cognitive behavioral principles-based treatment program — The treatment protocol had a total duration of 6 weeks. Two sessions were conducted each week, the first being a group session lasting 1.5 hours and the second an individual session lasting 45 minutes. During the group sessions, emotional disclosure and sharing of the experiences of patients with post COVID-19 syndrome were encouraged. During the individual sessions, a strong relationship was developed between the patient and the healthcare professional, with the healthcare professional helping the patient develop self-efficacy, thought monitoring, helpful self-talk, and reflection on changes in activity levels throughout the program.
  Arms: Cognitive behavioral principles-based treatment program group
Other: Control intervention — Patients received an informational brochure in a consultation with a health professional. The brochure explained the importance of physical activity to improve the health condition of these patients. Patients had the opportunity to ask any questions to the healthcare professional.
  Arms: Control group

SUMMARY:
Patients who have undergone COVID-19 infection often have long-term sequelae. One of the most prevalent sequelae is pain. The main objective of this research is to investigate the efficacy of a cognitive behavioral principles-based treatment program in fear avoidance beliefs, disability, pain catastrophizing and pain interference.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Agreed to participate.
* Post COVID-19 patients meeting the WHO definition for this disease.

Exclusion Criteria:

* Neurological or orthopaedic pathologies that limited voluntary movement.
* Cognitive impairment that prevented them from understanding and answering the questionnaires.
* Patients suffering from a reinfection with SARS-CoV-2.
* Patients who had been hospitalized due to COVID-19 infection.
* Patients who had pre-existing chronic pain according to the current IASP definition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Fear-avoidance belief changes | Baseline
  Fear avoidance beliefs will be assessed by the the Fear Avoidance Beliefs Questionnaire (FABQ). It consists of 16 sentences related to physical activity (first 5 items) and work (last 11 items).
Fear-avoidance belief changes | At 6 weeks at the end of the intervention
  Fear avoidance beliefs will be assessed by the the Fear Avoidance Beliefs Questionnaire (FABQ). It consists of 16 sentences related to physical activity (first 5 items) and work (last 11 items).

SECONDARY OUTCOMES:
Changes in functionality | Baseline
  Changes in functionality were measured using the World Health Organization Disability Assessment Schedule, WHODAS-2, which provides a global measure of disability and 7 domain-specific scores.
Changes in functionality | At 6 weeks at the end of the intervention
  Changes in functionality were measured using the World Health Organization Disability Assessment Schedule, WHODAS-2, which provides a global measure of disability and 7 domain-specific scores.
Changes in pain catastrophizing | Baseline
  Changes in pain catastrophizing were assessed with the pain catastrophizing scale. It consists of a 13-item scale with values from 0 to 4. The higher the score, the greater the pain catastrophization.
Changes in pain catastrophizing | At 6 weeks at the end of the intervention
  Changes in pain catastrophizing were assessed with the pain catastrophizing scale. It consists of a 13-item scale with values from 0 to 4. The higher the score, the greater the pain catastrophization.
Changes in pain interference | Baseline
  In the PROMIS PI, item category responses range from 1 to 5. T scores had a mean score of 50 and a standard deviation of 10 points. Low scores on the PROMIS PI represent less interference of pain with physical function, whereas high scores represent greater interference with physical function.
Changes in pain interference | At 6 weeks at the end of the intervention
  In the PROMIS PI, item category responses range from 1 to 5. T scores had a mean score of 50 and a standard deviation of 10 points. Low scores on the PROMIS PI represent less interference of pain with physical function, whereas high scores represent greater interference with physical function.
Changes in the sensory, affective and evaluative dimensions of pain. | Baseline
  The Short Form McGuill Pain Questionnaire (SF-MPQ) is a version of the original McGuill Pain Questionnaire, discovered by Melzak in 1987. This scale is divided into several parts. The first part consists of a list of 15 adjectives, including 11 sensory and 4 affective descriptors of pain (e.g., terrible, throbbing, etc.) on a scale ranging from 0 (none) to 3 (severe), giving an overall score ranging from 0 to 45, as well as two scores from 0 to 33 for the sensory subscale and 0 to 12 for the affective subscale. In addition, it includes a VAS scale that assesses the patient's pain in the last week. Finally, it includes a Present Pain Intensity Scale (PPI). The PPI is based on a single item measuring overall pain intensity. Patients are asked about their current level of pain on a 5-point Likert scale ranging from 0 (no pain) to 5 (unbearable). This scale has been shown to have excellent psychometric properties.
Changes in the sensory, affective and evaluative dimensions of pain. | At 6 weeks at the end of the intervention
  The Short Form McGuill Pain Questionnaire (SF-MPQ) is a version of the original McGuill Pain Questionnaire, discovered by Melzak in 1987. This scale is divided into several parts. The first part consists of a list of 15 adjectives, including 11 sensory and 4 affective descriptors of pain (e.g., terrible, throbbing, etc.) on a scale ranging from 0 (none) to 3 (severe), giving an overall score ranging from 0 to 45, as well as two scores from 0 to 33 for the sensory subscale and 0 to 12 for the affective subscale. In addition, it includes a VAS scale that assesses the patient's pain in the last week. Finally, it includes a Present Pain Intensity Scale (PPI). The PPI is based on a single item measuring overall pain intensity. Patients are asked about their current level of pain on a 5-point Likert scale ranging from 0 (no pain) to 5 (unbearable). This scale has been shown to have excellent psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada., Granada, Granada, Spain